CLINICAL TRIAL: NCT06755346
Title: The Acute and Chronic Effects of Cannabis on Reproductive Functions in Men
Brief Title: The Effects of Cannabis on Male Reproductive Functions
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kanako Hayashi (Other)
Collaborators: Washington State University (Other)
Responsible Party: Sponsor-Investigator, Kanako Hayashi, Professor, Washington State University
Organization: Washington State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: WSU_IRB#20730
Record Dates: First submitted 2024-12-19; First posted 2025-01-01 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Male Reproductive Problem
Keywords: Cannabis; Sperm counts and motility; Testosterone; Sperm epimutation
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol; nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cannabis users: non-vaping (No Intervention): Cannabis users (n=20) will be assigned to a non-vaping group.
- Cannabis users: placebo (Placebo Comparator): Cannabis users (n=20) will be assigned to a placebo group.
  Interventions: Drug: Cannabis (0%/ THC / 0% CBD)
- Cannabis users: 20mg THC in cannabis plant (Active Comparator): Cannabis users (n=20) will be assigned to a 20mg THC in cannabis group.
  Interventions: Drug: Cannabis plant (THC 20mg)
- Cannabis users: 40mg THC in cannabis plant (Active Comparator): Cannabis users (n=20) will be assigned to a 40mg THC group.
  Interventions: Drug: Cannabis plant (THC 40mg)
- non-cannabis users (No Intervention): Non-cannabis users (n=20) will be assigned to a non-vaping group.

INTERVENTIONS:
Drug: Cannabis plant (THC 20mg) — Cannabis flower - very High THC (>10%) / Low CBD (<1%)
  Other Names: marijuana
  Arms: Cannabis users: 20mg THC in cannabis plant
Drug: Cannabis (0%/ THC / 0% CBD) — THC (0%) / CBD (0%) - Placebo marijuana
  Arms: Cannabis users: placebo
Drug: Cannabis plant (THC 40mg) — Cannabis flower - very High THC (>10%) / Low CBD (<1%)
  Other Names: marijuana
  Arms: Cannabis users: 40mg THC in cannabis plant

SUMMARY:
The purpose of this study is to understand the direct effects of cannabis on male reproductive functions. The investigators plan to conduct a double-blind, placebo-controlled clinical trial to examine both the chronic and acute effects of cannabis use on male reproductive functions. Specifically, the investigators will examine the dose-dependent effects of acute cannabis use on male reproductive parameters, including sperm counts, motility, morphology, and testosterone levels, as well as sperm epimutations.

Participants [cannabis users will be randomly assigned to 1) non-vaping, 2) placebo (vaping without cannabis), and 2 doses of cannabis, 3) 20 and 4) 40mg of THC in cannabis flower obtained from the NIDA drug supply], and 5) non-cannabis users (naïve control, no cannabis or placebo exposure).

Participants will provide surveys (cannabis use and sexual functioning and satisfaction etc.), peripheral blood, and semen.

DETAILED DESCRIPTION:
The Volcano Vaporizer will be used to expose cannabis or placebo plants.

ELIGIBILITY:
Inclusion Criteria:

* Regular cannabis users (21~64 years-old men) who have used cannabis at least once a week for at least once a year or who have never used cannabis.
* Willingness to abstain from using cannabis on the day of the testing session (minimum 5 hours abstinence).

Exclusion Criteria:

* Women
* Adult men, 65 or older, and men under the age of 21
* Serious psychiatric conditions (e.g. psychosis, bipolar I and panic disorder)
* Family history of psychosis
* Chronic medical conditions (e.g., heart disease, diabetes)
* History of adverse experiences with cannabis (e.g., anxiety and panic attacks)
* Use of other illicit drugs (not cannabis) in the past 2 months
* Heavy alcohol use (>4 drinks, >4 times/week)
* Smoking/nicotine use
* Infrequent cannabis use (less than once a week for only cannabis users)
* BMI over 34
* Current use of corticosteroids and blood thinners

Ages: 21 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only biological men are eligible
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related sperm parameters | 30 minutes
  Sperm counts and motility, as well as DNA fragmentation, will be examined after vaping or no vaping.
Number of participants with treatment-related sperm epimutation | 30 minutes
  Differentially methylated regions in sperm will be analyzed to examine the effects of cannabis exposure.
Number of participants with treatment-related plasma testosterone and THC/THC metabolites | 4 hours
  Plasma testosterone and THC/THC metabolites will be analyzed to examine the effects of cannabis exposure.

SECONDARY OUTCOMES:
Number of participants with treatment-related stress reactivity and food intake | 4 hours
  After the vaping session and semen collection, participants will complete the Acute Stress Test. Plsama cortisol will be analyzed before and after the Acute Stress Test. During sobering (~4 hours), snacks (e.g., fruit snacks, granola bars, chips, chocolate, soda, juice, and water) will be available for participants. Investigators will monitor participants via the window in the adjacent room to monitor and record the snacks/beverages participants choose to consume.

CONTACTS AND LOCATIONS:
Overall Officials: Kanako Hayashi, PhD, Principal Investigator — Washington State University
Locations (1):
- Washington State University, Pullman, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is our first small study to obtain preliminary results. We plan to propose to investigate the effects of acute and chronic cannabis exposure on male reproductive functions in humans, which include single or multiple cannabis vaping exposures and multiple semen collections in the same individual with a larger sample of participants. The data from the large study will be shared.